CLINICAL TRIAL: NCT05367856
Title: Efficacy and Safety of Chidamide Combined With BEAM(Carmustine, Etoposide Cytarabine and Melphalan) Pretreatment in Autologous Transplantation for T-cell Lymphoma: a Single-center, Single-arm Clinical Study
Brief Title: Efficacy and Safety of Chidamide Combined With BEAM Pretreatment Regimen in Autologous Transplantation for T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chi-BEAM
Record Dates: First submitted 2022-04-25; First posted 2022-05-10 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: T Cell Lymphoma
Keywords: T cell lymphoma; Autologous Stem Cell Transplantation; Chidamide; BEAM
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chi-BEAM (Experimental): Patients in this arm will receive Chidamide Combined With BEAM(Carmustine, Etoposide Cytarabine and Melphalan) as Pretreatment Regimen of ASCT.
  Interventions: Drug: Chidamide combined with BEAM

INTERVENTIONS:
Drug: Chidamide combined with BEAM — Chidamide: 30mg po D-7,D-4,D-1 and D+3 Carmustine: 300mg/m2 ivgtt D-7 Etoposide: 100mg/m2/d ivgtt q12h D-6-D-3 Cytarabine: 200mg/m2/d ivgtt q12h D-6-D-3 Melphalan: 140mg/m2 ivgtt D-2

SUMMARY:
This single-center, single-arm clinical study will evaluate the efficacy and safety of Chidamide combined with BEAM Pretreatment Regimen in ASCT treatment of TCL patients.

DETAILED DESCRIPTION:
T cell lymphoma (TCL) is a group of highly heterogeneous aggressive non-Hodgkin lymphomas with different pathogenesis and clinical prognosis. Despite the survival benefits of Anthracycline-based chemotherapy bridging autologous stem cell transplantation (ASCT), 40% to 50% of TCL patients fail to respond to treatment and relapse or die within a short period of time. In 2021, a multicenter, single-arm, open Phase II trial of Chidamide combined with BEAC as a pretreatment regimen for ASCT of high-risk and relapsed/refractory lymphoma was presented at the ASH Meeting (NCT03629873). The results confirmed that Chidamide has a good prospect in ASCT. Chi-BEAC can increase 2Y-PFS from 55% to 93.3% and 2Y-OS from 58% to 94% in TCL patients after ASCT compared with the historical control group, with good tolerance.In order to provide a new program for improving survival rate, this single-center, single-arm clinical study will evaluate the efficacy and safety of Chidamide combined with BEAM Pretreatment Regimen in ASCT treatment of TCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. According to world Health Organization (WHO) classification of disease, T cell lymphoma (excepted IPI 0-1 point ALK+ anaplastic cell lymphoma) was confirmed by histology, CR or PR after first-line treatment;
2. 18≤ age ≤65 years old, male or female;
3. ECOG score 0-1;
4. No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) :

   * White blood cell count ≥3.0×109/L, absolute neutrophil count ≥1.5×109/L, Hemoglobin ≥90g/L, platelet ≥75×109/L;

     * Total bilirubin ≤1.5× upper normal value (ULN);

       * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× upper normal value (ULN);

         * Creatinine clearance was 44-133 mmol/L;
5. No cardiac dysfunction;
6. Life expectancy over 3 months;
7. The subject or his/her legal representative must provide written informed consent prior to conducting a special study examination or procedure.

Exclusion Criteria:

1. Central nervous system lymphoma was excluded;
2. Suffering from serious complications or severe infection;
3. A history of other malignant tumors within 5 years, excluding early tumors treated for curative purposes;
4. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.;
5. HBsAg, HCV or HIV positive. Positive HBV and HCV serology is allowed, but DNA/RNA testing must be negative;
6. Laboratory test value during screening;

   ① Neutrophils <1.5×109/L; Platelet <75×109/L;

   ② Bilirubin was 1.5 times higher than the normal upper limit, transaminase was 2.5 times higher than the normal upper limit;

   ③ The creatinine level is higher than 1.5 times the upper limit of normal value;
7. Left ventricular ejection fraction ≦ 50%;
8. Other concurrent and uncontrolled medical conditions considered by the investigator would affect the patient's participation in the study;
9. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol;
10. Pregnant or lactating women;
11. The researcher judged that the patients were not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of ASCT until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from an cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of ASCT to the date of death from any cause.
Complete remission rate | 3 months after the transplantation
  Percentage of participants with complete response was determined on 2014 Lugano criteria.
The time of hematopoietic reconstruction | 2 months after the transplantation
  The first day of neutrophils ≥0.5×109/L for 3 consecutive days was the time of successful implantation of granulocytes. Platelet ≥20.0×109/L for 7 consecutive days and the first day after platelet infusion was considered as the successful time of megakaryocytes implantation.
Transplantation-related adverse reactions | Baseline up to data cut-off (up to approximately 4 years)
  Transplantation-related adverse reactions are any untoward medical occurrence in a participant which is related to ASCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No